CLINICAL TRIAL: NCT05890079
Title: External Oblique Intercostal Plane Block for Postoperative Analgesia in Living Liver Donors
Brief Title: External Oblique Intercostal Plane Block for Liver Transplantation Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: anestezi2
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-05

CONDITIONS: Liver Transplantation; Donor; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcostal transversus abdominis plane block group (Active Comparator): The patients in subcostal transversus abdominis plane block group will be received subcostal transversus abdominis plane block and patient controlled analgesia with morphine for postoperative analgesia
  Interventions: Other: Subcostal transversus abdominis plane block
- External oblique intercostal plane block group (Active Comparator): The patients in External oblique intercostal plane block group will be received external oblique intercostal plane block and patient controlled analgesia with morphine for postoperative analgesia
  Interventions: Other: External oblique intercostal plane block

INTERVENTIONS:
Other: Subcostal transversus abdominis plane block — External oblique intercostal plane block will be administered at the end of the surgery and after skin closure.
  Arms: Subcostal transversus abdominis plane block group
Other: External oblique intercostal plane block — External oblique intercostal plane block will be administered at the end of the surgery and after skin closure. .
  Arms: External oblique intercostal plane block group

SUMMARY:
Postoperative pain management is one of the important factors to improve rehabilitation and enhance recovery. External oblique intercostal plane block may be used for abdominal wall analgesia to provide effective analgesia for abdominal surgery. The aim of this study is to investigate the postoperative analgesic efficacy of external oblique intercostal plane block and subcostal transversus abdominis plane block in living liver donors.

Researchers will compare the external oblique intercostal plane block group with subcostal transversus abdominis plane block to see if the external oblique intercostal plane block is effective for postoperative analgesia in living liver donors.

DETAILED DESCRIPTION:
Patients scheduled for living donor hepatectomy will be separated into 2 groups: Subcostal Transversus Abdominis Plane Block Group and External Oblique Intercostal Plane Block Group. Patients in Subcostal Transversus Abdominis Plane Block will be performed subcostal transversus plane block at the end of the surgery and after skin closure and received patient controlled analgesia with morphine for postoperative analgesia. Patients in External Oblique Intercostal Plane Block Group will be performed bilateral External Oblique Intercostal Plane Block at the end of the surgery and after skin closure and received patient controlled analgesia with morphine for postoperative analgesia. Morphine consumption for first postoperative 24 hours, visual analog scale scores, time to need for first rescue analgesia, amount of rescue analgesic drug, incidence of postoperative nausea and vomiting will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Patients with American Society of Anesthesiology (ASA) physical status I-II
* Patients scheduled for a living donor hepatectomy

Exclusion Criteria:

* Allergy to local anesthetics
* Coagulopathy
* Skin infection at the block area
* Advanced renal failure
* Chronic pain syndromes
* Alcohol or drug abuse
* Psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative 24 hours
  The amount of morphine required by the patient and given by the device will be recorded for the first 24 hours.

SECONDARY OUTCOMES:
Postoperative visual analog scale scores | Postoperative 24 hours
  Postoperative pain will be assessed using a visual analog scale (VAS) (from 0 = no pain to 10 = maximum possible pain) for the first 24 hours.
Rescue analgesic drug consumption | postoperative 24 hours
  The amount of rescue analgesic in mg required by the patient will be recorded for the first 24 hours.
Incidence of postoperative nausea and vomiting | postoperative 24 hours
  Number of patients developing postoperative nausea and vomiting will be recorded for the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Taylan Sahin, M.D., Principal Investigator — Istinye University
Locations (1):
- Istinye University Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Sahin T, Kavakli AS, Eren E, Aydin A, Sahin NK, Tokac M, Dinckan A. Ultrasound-guided external oblique intercostal plane block versus subcostal transversus abdominis plane block for postoperative analgesia in living liver donors: A prospective randomized trial. J Clin Anesth. 2025 Sep;106:111971. doi: 10.1016/j.jclinane.2025.111971. Epub 2025 Aug 19. PMID 40840080